CLINICAL TRIAL: NCT00930228
Title: Influence of Hyperandrogenemia on the Sleep-associated Slowing of Follicular LH Frequency in Adult Polycystic Ovary Syndrome
Brief Title: Effect of High Testosterone on Sleep-associated Slowing of Follicular Luteinizing Hormone (LH) Frequency in Polycystic Ovary Syndrome
Acronym: CRM004
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Chris McCartney, Associate Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 14067
Record Dates: First submitted 2009-06-24; First posted 2009-06-30 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Luteinizing hormone; Testosterone
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Flutamide

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Flutamide (Experimental): Flutamide 250 mg taken by mouth twice a day for 4 weeks. Flutamide is an androgen-receptor blocker.
  Interventions: Drug: Flutamide
- Placebo (Placebo Comparator): Placebo contains only inert ingredients and is not expected to exert any direct physiological effects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flutamide — Flutamide, 250 mg capsule for oral administration, twice a day for 4 weeks (or menstrual cycle length in normally-cycling controls)
  Other Names: Eulexin
  Arms: Flutamide
Drug: Placebo — Placebo, for oral administration, twice a day for 4 weeks (or menstrual cycle length in normally-cycling controls)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a testosterone receptor blocker (flutamide) will normalize sleep-wake luteinizing hormone pulse frequency relationships in women with polycystic ovary syndrome.

DETAILED DESCRIPTION:
During the follicular phase of the normal menstrual cycle, luteinizing hormone (LH) pulse frequency decreases during sleep. These decreases may be important to support follicle stimulating hormone (FSH) synthesis and secretion. Polycystic ovary syndrome (PCOS) is associated with a persistently rapid gonadotropin hormone-releasing hormone (GnRH) pulse frequency, an abnormality that may account for many of the hormonal manifestations of PCOS. Although one prior study suggests that nocturnal LH frequency decreases slightly in PCOS, methodological issues limit interpretation. Our preliminary data suggest that nocturnal LH frequency does not decrease in untreated PCOS, but that nocturnal decreases of LH frequency are restored with androgen receptor blockade (flutamide) in women with PCOS. We have two hypotheses: (1) Prior to flutamide administration, sleep-associated slowing of LH pulse frequency is less pronounced in women with PCOS compared to that of normally-cycling women in the late follicular phase of the menstrual cycle; (2) After 4 weeks of flutamide administration, sleep-associated LH frequency reduction in women with PCOS is similar to that of normally-cycling women in the late follicular phase of the menstrual cycle. Women with PCOS and normally-cycling women will be studied. For each study participant, LH pulse frequency will be determined (from 1500 to 0700 h) after 4 weeks of flutamide and after 4 weeks of placebo. Flutamide and placebo will be given in random order (i.e., cross-over study). Sleep will be formally evaluated. Flutamide will then be given for 4 weeks prior to reassessment of LH pulse frequency. LH pulse frequency will be analyzed by way of hierarchical mixed effect models. We will use statistical analyses to determine: (a) whether the wake vs. sleep difference in LH frequency is the same for PCOS and normal controls prior to flutamide, and (b) whether the mean wake vs. sleep difference in LH frequency is the same for the two groups after flutamide.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all participants:

* Subjects will be 18-35 years old; we use a cutoff age of 35 y because early menopause at this age is very rare.
* No significant health problems (other than PCOS and obesity).
* Subjects will be willing to strictly avoid pregnancy (using non-hormonal methods) during the time of study and must be willing and able to provide informed consent.

Inclusion criteria for normal controls:

* Controls will be healthy women with regular menstrual cycles and no evidence of hyperandrogenism.

Inclusion criteria for PCOS:

* PCOS will be defined according to NIH consensus criteria.

  * As such, subjects with PCOS will have hyperandrogenism, whether it is clinical (e.g., hirsutism) or biochemical (i.e., elevated plasma T).
  * Subjects with PCOS will also have oligo- or amenorrhea (i.e., < 7 periods per year) and no evidence for other endocrinopathies (e.g., hyperprolactinemia, Cushing's syndrome, etc.).

Exclusion Criteria:

* Being a study of GnRH pulse regulation in women with and without PCOS, men are excluded.
* Obesity associated with a diagnosed (genetic) syndrome, obesity related to medications (e.g., glucocorticoids), etc.
* Pregnancy or lactation.
* Virilization.
* A total testosterone > 150 ng/dl in women with PCOS (which suggests the possibility of a virilizing neoplasm) (confirmed on repeat).
* Elevated DHEAS (mild elevations may be seen in PCOS, and elevations < 1.5 times the upper limit of normal will be accepted in PCOS)(confirmed on repeat).
* Follicular 17-hydroxyprogesterone > 300 ng/dl, which suggests the possibility of congenital adrenal hyperplasia (if elevated during the luteal phase and there is a concern about the possibility of congenital adrenal hyperplasia, the 17-hydroxyprogesterone may be collected during the follicular phase, or >60 if oligomenorrheic).

  *NOTE: If a 17-hydroxyprogesterone > 300 ng/dl is confirmed on such repeat testing, an ACTH stimulated 17-hydroxyprogesterone < 1000 ng/dl will be required for study participation.
* A previous diagnosis of diabetes, a fasting glucose ≥ 126 mg/dl, or a hemoglobin A1c > 6.5%
* Abnormal TSH (subjects with adequately treated hypothyroidism, reflected by normal TSH values, will not be excluded; or, for a new diagnosis of hypothyroidism, further study will at the least be delayed pending appropriate treatment) (confirmed on repeat).
* Abnormal prolactin (mild elevations may be seen in PCOS, and elevations < 1.5 times the upper limit of normal will be accepted in this group) (confirmed on repeat).
* Evidence of Cushing's syndrome by history or physical exam.
* Hematocrit < 36% or hemoglobin < 12 g/dl (that is not reversed by iron treatment).
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; asthma requiring intermittent systemic corticosteroids; etc.)
* Liver test abnormalities (confirmed on repeat), with the exception that mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome.
* Abnormal sodium or potassium (confirmed on repeat); bicarbonate concentration <20 or >30 (confirmed on repeat); or elevated creatinine concentration (confirmed on repeat).
* Due to the amount of blood being drawn in the study, subjects with body weight < 110 lbs will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-01; Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Luteinizing hormone pulse frequency | One and two months

SECONDARY OUTCOMES:
Luteinizing hormone pulse amplitude | One and two months
Mean luteinizing hormone level | One and two months
Mean follicle stimulating hormone level | One and two months
Sleep study parameters | One and two months
  Sleep study parameters (sleep stage, overnight ventilatory variables) will be assessed when available

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have current plans to share IPD